CLINICAL TRIAL: NCT00859131
Title: Rabbit Anti-thymocyte Globulin Versus IL2 Receptor Antagonists in Combination With Tacrolimus, Corticosteroids and Mycophenolate Mofetil in a Predominantly High Risk Kidney Transplant Population.
Brief Title: Safety and Efficacy Study of Thymoglobulin Versus IL2 Receptor Antagonists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: thymo vs IL2
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2014-02

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — thymoglobulin; Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thymoglobulin (Active Comparator): Subjects receiving Thymoglobulin as induction agent in renal transplantation
  Interventions: Drug: Rabbit Antithymocyte globulin
- Zenapax (Active Comparator): subject who will receive daclizumab or basiliximab as induction agent in renal transplantation
  Interventions: Drug: Daclizumab

INTERVENTIONS:
Drug: Rabbit Antithymocyte globulin — 1.5 mg/kg IV pre-op, day 1, day 2, day 3, day 4
  Other Names: Thymoglobulin
  Arms: Thymoglobulin
Drug: Daclizumab — 1.0 mg/kg pre-op and 1.0 mg/kg on Day 7
  Other Names: daclizumab, zenapax
  Arms: Zenapax

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of induction therapy with Thymoglobulin in comparison with IL2 receptor antagonists (daclizumab or basiliximab).

DETAILED DESCRIPTION:
A 12 month, prospective, randomized, single center, open-label study to evaluate the safety and efficacy of Rabbit anti-thymocyte globulin versus IL2 receptor antagonists in combination with tacrolimus, corticosteroids and mycophenolate mofetil in a predominantly high risk kidney transplant population.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 75 years of age
* Male or female patients who are primary or repeat cadaveric, living unrelated or non- Human leukocyte antigen (HLA) identical living related donor renal transplant recipients
* Female patients of child bearing potential must have a negative urine or serum pregnancy test within the past 48 hours prior to study inclusion.
* The patient has given written informed consent to participate in the study

Exclusion Criteria:

* Patient has previously received or is receiving an organ transplant other than a kidney.
* Patients who are recipients of a multiple organ transplant.
* Patient has received a primary or re-transplant from an HLA-identical living donor.
* Any positive cross-match.
* Patient is the recipient of a pediatric donor kidney from a pediatric donor aged 8 years or less.
* Patient has received an ABO incompatible donor kidney.
* Recipient or donor is known to be seropositive for hepatitis C virus (HCV) or B virus (HBV) except for hepatitis B surface antibody positive.
* Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV).
* Patient has uncontrolled concomitant infection or any other unstable medical condition that could interfere with the study objectives.
* Patients with thrombocytopenia (<75,000/mm3 ), with an absolute neutrophil count of < 1,000/mm3); and/or leucopoenia (< 2,000/mm3), or anemia (hemoglobin < 6 g/dL) prior to study inclusion.
* Patient is taking or has been taking an investigational drug in the 30 days prior to transplant.
* Patient has a known hypersensitivity to tacrolimus, mycophenolate mofetil, rabbit anti-thymocyte globulin, daclizumab or corticosteroids.
* Patients with severe diarrhea or other gastrointestinal disorders that might interfere with their ability to absorb oral medication.
* Patients with a history of malignancy within the last five years, except for successfully excised squamous or basal cell carcinoma of the skin.
* Patient is pregnant or lactating, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by positive human Chorionic Gonadotropin (hCG) laboratory test.
* Women of childbearing potential must use two reliable forms of contraception simultaneously, unless they are status post bilateral tubal ligation, bilateral oophorectomy, or hysterectomy. Effective contraception must be used before beginning study drug therapy, for the duration of the study and for 6 weeks following completion of the study.
* Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator.
* Inability to cooperate or communicate with the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Chavin, MD,PhD, Study Chair — Medical University of South Carolina; Nicole Pilch, PharmD, Study Chair — Medical University of South Carolina; David Taber, PharmD, Study Chair — Medical University of South Carolina; Prabhakar Baliga, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Palanisamy AP, Al Manasra AR, Pilch NA, Dowden JE, Nadig SN, McGillicuddy JW, Baliga PK, Chavin KD, Taber DJ. Induction therapy: clinical and quality of life outcomes in aged renal transplant recipients. Clin Transplant. 2015 Mar;29(3):222-6. doi: 10.1111/ctr.12507. Epub 2015 Jan 27. PMID 25557762
- [Derived] Pilch NA, Taber DJ, Moussa O, Thomas B, Denmark S, Meadows HB, McGillicuddy JW, Srinivas TR, Baliga PK, Chavin KD. Prospective randomized controlled trial of rabbit antithymocyte globulin compared with IL-2 receptor antagonist induction therapy in kidney transplantation. Ann Surg. 2014 May;259(5):888-93. doi: 10.1097/SLA.0000000000000496. PMID 24513787

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thymoglobulin | Zenapax
Started | 102 | 98
Completed | 102 | 98
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thymoglobulin | Zenapax | Total
Number analyzed (Participants) | 102 | 98 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (13) | 49 (14) | 50.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 36 | 79
  Male | 59 | 62 | 121

OUTCOME MEASURES:

1. Primary Outcome: Treatment Efficacy Will be Defined as the Number of Patients With Biopsy Proven Acute Rejection at One Year Post-transplant.
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Thymoglobulin | Zenapax
Number analyzed (Participants) | 102 | 98
participants | 6 | 10

2. Secondary Outcome: Number of Patients Requiring Antilymphocyte Therapy for Acute Rejection.
Time Frame: One year
Measure: Number; unit: Patients
Arm/Group | Thymoglobulin | Zenapax
Number analyzed (Participants) | 102 | 98
Patients | 3 | 8

3. Secondary Outcome: Graft Survival at One Year Post-transplant
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Thymoglobulin | Zenapax
Number analyzed (Participants) | 102 | 98
participants | 101 | 95

4. Secondary Outcome: Incidence of Post-transplant Infections, Including, But Not Limited to, CMV Infection and Disease, BK Infection and Nephropathy, Other Opportunistic Infections, Urinary Tract Infections, Pneumonia, and Sepsis
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | Thymoglobulin | Zenapax
Number analyzed (Participants) | 102 | 98
participants | 52 | 58

5. Secondary Outcome: Incidence of Post-transplant Malignancies, Including Post-transplant Lymphoproliferative Disease (PTLD) and Skin Cancers.
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Thymoglobulin | Zenapax
Number analyzed (Participants) | 102 | 98
participants | 3 | 0

6. Secondary Outcome: Incidence of Leukopenia, Defined as a Total White Blood Cell Count of Less Than 2,000 Cells/mm3
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Thymoglobulin | Zenapax
Number analyzed (Participants) | 102 | 98
participants | 21 | 4

7. Secondary Outcome: Incidence of Thrombocytopenia, Defined as a Platelet Count of Less Than 100,000 Cells/mm3
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Thymoglobulin | Zenapax
Number analyzed (Participants) | 102 | 98
participants | 43 | 13

ADVERSE EVENTS:
Arm/Group | Thymoglobulin | Zenapax
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/98
Other Adverse Events (participants affected / at risk) | 37/102 | 44/98
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Thymoglobulin (N=102) | Zenapax (N=98)
BK Viremia (Blood and lymphatic system disorders) | 13 | 19
CMV (Immune system disorders) | 29 | 18
Bacterial Infection (Infections and infestations) | 10 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No